CLINICAL TRIAL: NCT04561713
Title: Development of a Virtual Reality Application for the Diagnosis of Childhood ADHD: an Exploratory Study
Brief Title: Virtual Reality and Diagnostic of Attention Deficit Hyperactivity Disorder (ADHD) (PADA1)
Acronym: PADA1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/33
Record Dates: First submitted 2020-08-03; First posted 2020-09-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Virtual reality
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Deficit Hyperactivity Disorder (ADHD) (Experimental): Children aged 8 to 12 diagnosed with ADHD
  Interventions: Procedure: Virtual reality task
- Control (Sham Comparator): Control group of healthy ADHD children matched in age, gender and laterality to children in ADHD group
  Interventions: Procedure: Virtual reality task

INTERVENTIONS:
Procedure: Virtual reality task — Virtual reality application in an immersive room (CAVE) in three dimensions to assess child's sustained attention in a dynamic environment that is as close as possible to everyday situations.

SUMMARY:
The aim of this study is to develop an application in order to identify the most relevant cognitive and behavioral parameters for the diagnosis of Attention Deficit Hyperactivity Disorder (ADHD) in conditions closer to reality

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) is the most common neurodevelopmental disorder in school-aged children. This disorder is characterized by a symptomatic triad associating, inattention, hyperactivity and impulsivity. Cognitive, emotional and behavioral dysfunctions have a strong impact on the school, family and social domains of the child. The clinical diagnosis of ADHD is all the more difficult because there are currently no biological, clinical or psychological markers that accurately measure the symptoms of ADHD. The diagnosis is made during interviews with specialist doctors allowing the collection of information from parents and the child. Virtual reality technology is most recognized as a tool for assessment, rehabilitation of cognitive processes and functional skills. In addition to traditional diagnostic assessment methods, a virtual reality application in an immersive room (CAVE) in three dimensions could objectively assess the child in a dynamic environment that is as close as possible to everyday situations

ELIGIBILITY:
Inclusion Criteria:

Group of children with ADHD :

* Children aged 8 to 12 diagnosed with ADHD (according to DSM-V criteria)
* Positive ADHD diagnosis with standardized maintenance of Kiddie-Sads
* Naïve drug treatment for ADHD
* Schooled in a classic environment
* Intellectual Quotient> 80 (4 subtests of WASI, or WISC IV-R / WISC-V less than 2 years old)
* Having French as mother tongue
* Children benefiting from a social security scheme
* Signing of free, informed and written consent by the child and the holders of parental authority Group of children controls

Children aged 8 to 12 years undiagnosed ADHD (according to DSM-V criteria) :

* Not presenting with ADHD at standardized maintenance Kiddie-Sads
* Schooled in a classic environment
* Intellectual Quotient> 80 (4 subtests of WASI)
* Having French as mother tongue
* Children benefiting from a social security scheme
* Signing of free, informed and written consent by the child and the holders of parental authority

Exclusion Criteria:

* Positive diagnosis with standardized maintenance of Kiddie-Sads for the following disorders: mood disorders, psychotic disorders, autism spectrum disorders, severe anxiety disorders and severe tic disorders
* Presenting a hearing or vision diagnosis diagnosed that does not allow the task to be performed in virtual reality
* Neurological disorders
* Photosensitive Epilepsy (contraindication to immersion in virtual reality)
* Treatment with psychostimulants or other psychotropic drugs
* Unable to complete the virtual reality task during the familiarization session

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Average number of commission errors | From one day to 8 weeks after day 0
  Average number of commission errors to the virtual reality task

SECONDARY OUTCOMES:
Average reaction time (ms) | From one day to 8 weeks after day 0
  The average reaction time (ms) to the virtual reality task
Average number of omission errors | From one day to 8 weeks after day 0
  Average number of omission errors to the virtual reality task
Average number of head movement | From one day to 8 weeks after day 0
  The average amount of head movement to the virtual reality task
Average number of foot movement | From one day to 8 weeks after day 0
  The average amount of foot movement to the virtual reality task
Percentage | From one day to 8 weeks after day 0
  The percentage of periods with emotions during the virtual reality task
Percentage of period with presence of Emotion | From one day to 8 weeks after day 0
  Percentage of period with presence of Emotion (Engagement > 50) during the task of virtual reality (range from 0 to 100).
Mean Emotion intensity (Engagement) | From one day to 8 weeks after day 0
  Mean Emotion intensity (Engagement) during the task of virtual reality (range from 0 to 100).
Mean Emotion valence | From one day to 8 weeks after day 0
  Mean Emotion valence (negative or positive emotion) during the task of virtual reality (range from -100 to 100).
Average reaction time (ms) | Day 0
  The average reaction time (ms) to the Continuous Performance Test (CPT) wich is a neuropsychological assessment test of sustained attention
Average number of commission errors | Day 0
  The average number of commission errors to the CPT neuropsychological task
Average number of omission errors | Day 0
  The average number of omission errors to the CPT neuropsychological task
Total score with the Attention-Deficit Hyperactivity Disorder-Rating Scale. | Day 0
  Scale to assess the severity of the 18 symptoms of DSM related to ADHD, the higher score mean a worse outcome. Max value : 54
Inattention score with the Attention-Deficit Hyperactivity Disorder-Rating Scale | Day 0
  Inattention score with the Attention-Deficit Hyperactivity Disorder-Rating Scale. With inattention (items impairs) max value = 27, the higher score mean a worse outcome
Hyperactivity score with the Attention-Deficit Hyperactivity Disorder-Rating Scale | Day 0
  Hyperactivity score with the Attention-Deficit Hyperactivity Disorder-Rating Scale. Hyperactivity (items pairs) max value=27, the higher score mean a worse outcome
Executive Performance Inventory Score | Day 0
  Executive Performance Inventory Score with Behavior Rating Inventory of Executive Function (BRIEF) questionnaire. Min value=30 and max value=100 the higher score mean a worse outcome.
Quality of life (VSPA-e) score | Day 0
  Quality of life score with VSPA-e questionnaire. Min value= 0 and max value=100 the higher score mean a worse outcome
Quality of life (KIDSCREEN) score | Day 0
  Quality of life with KIDSCREEN questionnaire. Min value= 0 and max value=100 the higher score mean a better outcome.
Acceptability score of virtual reality tool | From one day to 8 weeks after day 0
  Acceptability score of virtual reality tool. Min value= 6 and max value=30 the higher score mean a better outcome.
Acceptability score of classic neuropsychological test | From one day to 8 weeks after day 0
  Acceptability score of classic neuropsychological test. Min value= 6 and max value=30 the higher score mean a better outcome.
Simulator Sickness score | From one day to 8 weeks after day 0
  Score on the "Simulator Sickness" questionnaire. Min value= 0 and max value=63 the higher score mean a worse outcome.
Feeling of presence score | From one day to 8 weeks after day 0
  Score at the "feeling of presence" scale. Min value= -42 and max value=+42 The higher score mean a better immersion.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Arthur MICOULAUD-FRANCHI, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France